CLINICAL TRIAL: NCT05394428
Title: Novel Functional Anatomic and Biomarker Indices of Radiation-Induced Female Sexual Toxicities in a Multi-Center Cohort
Brief Title: A Multi Center Study of Sexual Toxicities After Radiotherapy
Acronym: STAR
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Emory University (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Deborah Marshall, Principal Investigator, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 20-2369
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Malignant Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood Samples; Microbiome Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with female sexual organs treated with pelvic radiotherapy: Patients with female sexual organs treated with pelvic radiotherapy.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this research is to understand how radiotherapy and other cancer treatments impact sexual function in female cancer patients and to try to answer a question about why some patients who receive radiotherapy are more likely to have side effects than others. The results of this study may improve our understanding of why sexual side effects occur and in turn develop predictive models and biomarkers of sexual side effects and other side effects that may impact sexual function. The results of this study may also lead to improvements in the techniques used to deliver radiotherapy or the development of interventions that will prevent or reduce sexual side effects and improve quality of life for female patients with cancer.

DETAILED DESCRIPTION:
Participants will be asked too:

* Give consent for past and future access to medical record information. At each timepoint, the study team will collect data from electronic medical record about (demographics), health conditions and treatments, studies (labs, imaging) and outcomes (response to treatment and toxicity).
* Quality of Life/Toxicity Questionnaires (Cohort: STAR*QOL): The study staff will administer (in clinic, by phone, or by email) health and quality of life/toxicity questionnaires that will ask questions about general well-being and side effects from treatment, which will take approximately fifteen minutes each time. These questionnaires are required to participate in the study. The questionnaires will be completed before treatment, after treatment, then every six months for two years. In addition, the study team would like participants to complete a questionnaire every year thereafter and will continue to ask participants to complete the questionnaires as long as they are enrolled, unless they decide no longer to participate.
* Blood Sample Collection (Cohort: STAR*QOL): a small amount of blood will be drawn from participants arm (one specimen up to 45 mL or about 3 tablespoons). The blood may be drawn at the same time as routine blood draw for medical care, as part of their participation in another research study, or solely for this study. Biological blood samples will be collected by the treatment team before treatment, at the end of treatment, 5 weeks after treatment and every 6 months thereafter for two years. Participants may be asked if they would like to continue annually after 2 years.
* Microbiome Sample Collection (Cohort: STAR*QOL): If participants choose to participate, biological microbiome samples (a vaginal and stool sample) will be collected at home using a home collection kit before treatment, after treatment and annually for two years.Participants may be asked if they would like to continue annually thereafter.

The research on biospecimens may include whole genome sequencing (determining the order of DNA building blocks (nucleotides) in their genetic code) and other studies on the DNA such as how DNA is modified or turned in to proteins.

Ultrasound Imaging (Cohort: STAR*Biomarker):

If participants choose to participate, ultrasound images will be collected by the treatment team before treatment, after treatment and every 6 months for two years thereafter, and can be performed at their scheduled office visit for their cancer care rather than requiring an additional visit. Additional imaging time may also be added onto their standard MRI scans to allow for additional images to be captured. Participants may be asked if they would like to continue annually after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with female sexual organs ages 18 and older.
* Patients must meet at least one of the following two criteria:

  * have been sexually active in the 36 months prior to initiating cancer treatment.
  * have the intent to be sexually active in the 24 months following treatment..
* Patients must be able to provide consent and be willing to participate.
* Patients must have primary anal, rectal, cervical, uterine, vaginal, or vulvar cancer planned to receive pelvic radiotherapy.** Patients must have an Eastern Cooperative Oncology Group performance status <=2.

Exclusion Criteria:

* planned for or undergone extensive pelvic surgery (e.g. pelvic exenteration, non-TME techniques, or surgeries otherwise affecting pudendal neurovasculature);
* have clinically or radiologically detectable widespread metastasis;
* have limited life expectancy due to comorbid disease;
* have a personal history of cancer other than non-melanoma skin cancer in the last 5 years;
* have contraindications or strong relative contraindications to radiotherapy at baseline as determined by the treating radiation oncologist (pregnancy, lactation, genetic susceptibility to cancer from ionizing radiotherapy, connective tissue disorders, inflammatory/irritable bowel disease, history of prior pelvic radiotherapy).
* have persistent, infectious gastroenteritis, colitis or gastritis;
* have persistent or chronic diarrhea of unknown etiology; have recurrent or untreated GI infection (clostridium difficile or H. pylori);
* have current or recurrent vaginal infection;
* have current or recent antibiotic use (within 2 months).

Patients may be enrolled regardless of previous local or systemic treatments received prior to enrollment in the STAR Study.

Patients may be enrolled on the STAR Study concurrently with another study or clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a study of female sexual organs, therefore patients of any gender identity with female sexual organs can participate.
Study Population: Adult female patients treated with pelvic radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Establish Sexual Quality of Life Cohort | 2 years
  Establish a cohort of patients with female sexual organs receiving radiotherapy

SECONDARY OUTCOMES:
Describe sexual quality of life | 2 years
  Describe sexual quality of life for patients with female sexual organs receiving radiotherapy
Describe dosimetric predictors of sexual outcomes | 2 years
  Describe the dosimetric predictors of sexual outcomes for patients with female sexual organs receiving radiotherapy
Describe imaging predictors of sexual outcomes | 2 years
  Describe the imaging predictors of sexual outcomes for patients with female sexual organs receiving radiotherapy
Describe microbiome predictors of sexual outcomes | 2 years
  Describe the microbiome predictors of sexual outcomes for patients with female sexual organs receiving radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Deborah C Marshall, MD MAS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported including individual-level quality-controlled individual microbiome 16s rRNA genomic sequencing and clinical correlative information.
  Data repositories will include an institutional controlled-access database available to the investigators and any other qualified investigator who has sought the approval of the investigators to pursue additional studies, in addition to depositing the study data in the unrestricted-access Sequence Read Archive database, a NIH-designated Data Repository supported by the NCBI.
Supporting Information: CSR
Time Frame: Data will be submitted approximately 3 months after the data have been generated, following data cleaning and quality control, and released within 6 months.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose for institutional controlled access data.
  Unrestricted access anonymized data are available indefinitely at (Link to be included in the URL field below).
URL: https://trace.ncbi.nlm.nih.gov/Traces/sra/